CLINICAL TRIAL: NCT01591109
Title: A Reversal in the Vascularity of Metastatic Liver Tumors in Patients With Colorectal Cancer After the Cessation of Anti-VEGF Therapy: A Study Using Contrast-enhanced Ultrasonography and Histological Techniques.
Brief Title: A Reversal in the Vascularity of Metastatic Liver Tumors From Colorectal Cancer After the Cessation of Anti-VEGF Therapy
Status: Completed | Type: Observational
Sponsor: NHO - Matsumoto Medical Center (Other Government)
Responsible Party: Principal Investigator, Hiroshi Kitamura, Chief of Surgical Department, NHO - Matsumoto Medical Center
Other Study IDs: 24-1
Record Dates: First submitted 2012-05-02; First posted 2012-05-03 (Estimated); Last update posted 2012-05-03 (Estimated); Status verified 2012-05

CONDITIONS: Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Time Perspective: Retrospective
Biospecimen Retention: Samples Without DNA — formalin fixed oarafin embedded block of liver specimen
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Bevacizumab including chemotherapy: Patients treated with bevacizumab including chemotherapy for metastatic liver tumor derived from colorectal cancer before metastasectomy.
- no adjuvant chemotherapy: Patients with no adjuvant chemotherapy including bevacizumab

SUMMARY:
Objective: To assess the effect of bevacizumab on tumor vessels, and the reversibility of the effect, using contrast-enhanced ultrasonography (CEUS) and histology in patients with metastatic liver tumors derived from colorectal cancer.

Background Data: Direct evidence on the reversibility of any change in tumor vascularity upon bevacizumab cessation in the clinical setting is lacking.

Methods: The study included 10 patients who received chemotherapy including bevacizumab, experienced a reduction in tumor vascularity as demonstrated by CEUS and consequently underwent liver resection. CEUS was performed before and immediately after 4 courses of chemotherapy and one day before surgery. The number of microvessels highlighted by anti-CD34 antibody in the viable tumor tissue was counted to quantify the microvessel density (MVD). As a control, 10 surgical specimens from 10 patients who had not received chemotherapy were examined.

ELIGIBILITY:
Inclusion Criteria:

* patients who received chemotherapy (FOLFOX) including bevacizumab. The patients had an associated reduction in tumor vascularity as estimated by ultrasonography and consequently underwent surgical resection of the metastatic liver tumors for curative purposes.

Exclusion Criteria:

* none

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Residents cared by the institution this study was perfomed.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2010-01; Primary Completion 2012-04 (Actual); Study Completion 2012-04 (Actual)